CLINICAL TRIAL: NCT05885971
Title: Detection of Eating Disorders in Pregnant Women
Acronym: PREGN'ED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-A00529-36
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Eating Disorders; Pregnancy Related
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of pregnant women with eating disorder (Other)
  Interventions: Diagnostic Test: Administration of the SCOFF-F and EDE-Q questionnaires
- Group of pregnant women with no eating disorder (Other)
  Interventions: Diagnostic Test: Administration of the SCOFF-F and EDE-Q questionnaires

INTERVENTIONS:
Diagnostic Test: Administration of the SCOFF-F and EDE-Q questionnaires — The participants will answer to the SCOFF-F and EDE-Q questionnaires as well as socio-demographic questions

SUMMARY:
Eating disorders (ED) are insufficiently detected and belatedly or not treated during pregnancy.

There are many screening questionnaires for eating disorders in the literature, but we note the absence of a specific and validated tool for their screening during pregnancy, which would make it possible to differentiate maternal dietary concerns related to pregnancy from symptoms linked to a proven eating disorder.

The main objective of the study is to evaluate which items of the Sick Control One stone Fat Food (SCOFF-F) and Eating disorders examination questionnaire (EDE-Q) questionnaires could be specific to an ED during pregnancy and not related to the simple state of pregnancy, by comparing the answers of pregnant women, for whom the diagnosis of ED has been made, to those of pregnant women without an ED.

ELIGIBILITY:
Inclusion Criteria:

* Adult pregnant woman
* Woman with current diagnosed Eating Disorders or without Eating Disorders
* Having a good command of the French language
* Having given their consent for their participation in the research

Exclusion Criteria:

* Underage pregnant woman
* Woman who does not have a good command of the French language.
* Woman with past Eating Disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Specific Eating Disorders items in pregnant women | 36 months
  A discriminant factor analysis will be used to study whether there are elements that can distinguish women with an Eating Disorders from those who do not have one during pregnancy.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Henri Laborit, Poitiers, France